CLINICAL TRIAL: NCT01987024
Title: Advantage of Detection of phIGFBP-1 to Reduce Hospitalization Time for Stable Patients With a Risk of Preterm Labour.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-A00780-45; 2013-21 (Other: AP HM)
Record Dates: First submitted 2013-09-16; First posted 2013-11-19 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Patients With a Risk of Preterm Labour

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group A-usual procedure (Active Comparator)
  Interventions: Other: usual procedure
- groupB- actim partus (Experimental)
  Interventions: Device: Actim Partus® test

INTERVENTIONS:
Device: Actim Partus® test
  Arms: groupB- actim partus
Other: usual procedure
  Arms: group A-usual procedure

SUMMARY:
It consists of evaluating the advantage of routine detection of phIGFBP-1 to reduce the total duration of hospitalization for patients with a risk of preterm labor before 32 weeks of gestation without increasing the number of preterm labour.

Methods Patient with a risk of preterm labor (ultrasound cervical length < 25 mm +/- described or recorded uterine contractions) before 32 weeks of gestation will be hospitalized to receive tocolytic drugs and antenatal corticosteroid therapy according to our gold standard protocol. After 48 hours, they will be assessed by examination, external tocodynamometry and the measure of cervical length by ultrasound. Stabilized patients will be included and randomized into 2 groups of 210 patients each. The first group "A" will benefit from the standard protocol (extended hospitalization of 2 or 4 days according to the clinical and ultrasound assessment); whereas the second group, "B", will have the benefit of the detection of phIGFBP-1.If the result proves negative, patients could be discharged early at day 2. In the case of a positive result, patients will follow the standard procedure because of the low positive predictive value of the test. The main outcome is the total duration of hospitalization.

Study duration The trial period will be 36 months.

Expected results The use of detection of IGFBP-1 would enable us to select patients at risk and to decrease the duration of hospitalization in the case of a negative result.

Perspectives The negative predictive value of phIGFBP-1 test could be useful to select patients with stabilized risk of preterm labor, who could be discharged early. Moreover it could be used, in the Perinat Sud network, to decide if patients with a risk of preterm labor would benefit from hospitalization in a level II or III maternity ward.

ELIGIBILITY:
Inclusion Criteria:

* • Women aged 18 years or more,

  * Women with a single intrauterine pregnancy with a term consistent with the LMP and / or ultrasound of the first quarter,
  * Women with a pregnancy in which the term is greater than 24 weeks and strictly less than 34 weeks,
  * initially consultant Woman (D0):
* For painful uterine contractions associated with ultrasound measurement of a neck (LC) of less than 25 mm,
* Or cervical changes discovered incidentally during a vaginal examination confirmed by LC <25 mm,
* Or during a routine ultrasound with LC <25 mm;
* Patient with a MAP stabilized in terms Clinical Ultrasound in D2:

Clinical criteria: absence of painful uterine contractions described or strictly less than 3 uterine contractions recorded during an external électrocardiotocographie for 30 minutes; And sonographic criteria: cervicométrie measured steady J2 (+ / - 10%) or increased relative to the cervicométrie J0.

- Women who have signed a written informed consent.

Exclusion Criteria:

* - Minor Female,
* Women with a multiple pregnancy,
* Women with a pathological whose late intrauterine growth preeclampsia, fetal malformations, maternal-fetal immunizations, abnormal amount of amniotic fluid (polyhydramnios / oligohydramnios), abnormal insertion of pregnancy placenta (low inserted / previa acreta / percreta)
* Women with pregnancy circled,
* Women with premature rupture of membranes or signs of chorioamnionitis,
* Women with bleeding irregularities,
* Women with uterine malformation (septate uterus, bicornuate, polyfibromateux)
* Women are not affiliated with the social security system,
* Women who can not receive an informed information
* Women who have not signed the informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2013-10; Primary Completion 2019-09-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
vaginal cervical sampling | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France